CLINICAL TRIAL: NCT04024111
Title: The Development and Evaluation of a Social Skills Group Training for Australian Children on the Autism Spectrum
Brief Title: Social Groups for Australian Children on the Autism Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Curtin University (Other)
Collaborators: Autism Association of Western Australia (Unknown); Stan Perron charitable trust (Unknown); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sonya Girdler, Professor, Curtin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRE2017-0245-34
Record Dates: First submitted 2019-07-12; First posted 2019-07-18 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Social groups; Active contol group; Children; Australian
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated into an intervention group (KONTAKT Australia) and an active control group (Social Art group).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The Assessor is blind to the participant's allocation to the intervention and active control group and the participants and carers are told they are participating in different social groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KONTAKT(c) (Experimental): A social skills group training
  Interventions: Behavioral: KONTAKT(c)
- Art group (Active Comparator): A social Art group
  Interventions: Other: Art group

INTERVENTIONS:
Behavioral: KONTAKT(c) — KONTAKT is a manualized Social skills group training program designed for children and adolescents on the Autism Spectrum aimed at improving communication, social interaction skills, the severity of ASD symptoms, and the ability to empathise and adapt in a group setting. The KONTAKT participants (4-8 participants) meet face to face weekly for 16 weeks for 75 minutes facilitated by two health professionals with experience of running groups for autistic children
  Arms: KONTAKT(c)
Other: Art group — Art program, a manualized Art group delivered in a social format, has been designed for children on the Autism Spectrum delivered by health professionals with experience of running social groups for Autistic children. The Art program's participants (4-8 participants) meet face to face weekly for 16 weeks for 75 minutes.
  Arms: Art group

SUMMARY:
This study evaluates the KONTAKT social skills group training in Australian children on the autism spectrum compared to an active control group which is a group Art class

DETAILED DESCRIPTION:
KONTAKT is a manualized Social Skills Group Training program designed for children and adolescents with ASD which aims to improve communication, social interaction skills, reduce the severity of ASD symptoms, improve the ability to empathise and adapt in a group setting. A large randomized controlled trial in Sweden found that adolescents who participated in KONTAKT demonstrated improvements in social skills, behaviour, reduced stress and improved overall functioning as reported by parents immediately following and at three months after the program. However, social skills are at least in part influenced by social cultural contexts and there is a need to understand the feasibility, acceptability and effectiveness of KONTAKT in an Australian context. Moreover, in the previous studies, the social skills groups were compared to treatment as usual groups. Therefore, this study evaluates the KONTAKT social skills group training in Australian children on the autism spectrum compared to an active control group which is a group art class

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 8 to 12
* Clinical consensus diagnosis of ASD as defined by DSM-5 and confirmed by the Autism Diagnostic Observation schedule-2
* IQ scores > 70 as measured by the Wechsler Abbreviated Scale of Intelligence - Second Edition (WASI-II)

Exclusion Criteria:

* Existing prior comorbid externalizing behaviours as assessed by the Childhood Behaviour Checklist (CBCL).
* Clinically assessed self-injurious behaviour • Low intrinsic motivation to participate in a social skills training group
* Insufficient English language skills

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in the Goal Attainment Scale (GAS) | Baseline (week 0), Post-test (week 20) and follow up (week 36) and long follow up (74 weeks)
  The GOAL Attainment Scale will be used to measure if the participants have achieved the goals they have set for the program. Using the scale the children's primary outcome. Using the scale the participants personally meaningful social goals will be specified, and a behavioural expectation that ranges from the worst to the best possible outcome will be listed for each goal. This allows qualitative data to be quantified in relation to the success of the participant in achieving expectations of change. The achievement of these goals will be scored via the GAS scoring system of "-2" showing the participant's current level of performance, "-1" less than expected, "0" the expected progress, and "+1" and "+2" indicative of progress above the expected level
Change in Social Skills Assessment Questionnaire (SSAQ) | Baseline (week 0), Post-test (week 20) and follow up (week 36) and long follow up (74 weeks)
  Social Skills Assessment Questionnaire (SSAQ), is a 23-item parent proxy questionnaire measuring the change in a child's social skills abilities. the measure is rated on a 3-point Likert scale from "worse than peers" to "Better than peers". Higher total scores show better outcome. This measure has been used with the ASD population before.

SECONDARY OUTCOMES:
Change in the Emotion Regulation Checklist (ERC) | Baseline (week 0), Post-test (week 20) and follow up (week 36) and long follow up (74 weeks)
  2.3. The parents will fill this questionnaire (Parent form). This is a 24-item measure assessing : negativity/lability and emotion regulation. The questionnaire is designed to measure represents a different aspect of emotionality from a strengths perspective, i.e. emotional intelligence, resilience and coping and social and emotional competence. Responses are rated on a 4-point Likert scale, ranging from "rarely" to "almost".
Change in the Negative Incidents and Effects of Psychological Treatment (NEQ) | Post-test (week 20)
  The parents (parent proxy) will fill this questionnaire. The NEQ is a 32-item questionnaire requiring adolescents to quantify, on 5-point Likert scale with response options ranging from "Not at all" to "Extremely", any negative events experienced during the intervention period, asking participants to attribute their causality to either the program or external circumstances
Change in the Child Health Utility 9D (CHU9D) | Baseline (week 0), Post-test (week 20) and follow up (week 36) and long follow up (74 weeks)
  The children will fill this questionnaire. This is a 9-dimension Health related quality of life scale (worried, sad, pain, tired, annoyed, school work, sleep, daily routines and activities), designed to estimate the adolescent's Quality adjusted life years (QALY), providing a standardized measure of disease burden. The measure is rated on a 5-point scale with a "don't" sentence linked with no problems (e.g. I don't feel sad today) and "very" with the participant experiencing a lot of problems (e.g. I feel very sad). Calculation of an universal score is supported by an adolescent specific scoring algorithm, with 1 representing 'full health' and 0 'death'.
Change in Treatment Inventory of Costs in Patients (TIC-P) | Baseline (week 0), Post-test (week 20) and follow up (week 36) and long follow up (74 weeks)
  The parents will fill this questionnaire (Parent form). This will be measured via a tailored version of the Trimbos/iMTA questionnaire for patients with a psychiatric disorder (TiC-P), a well-established questionnaire examining health care usage as well as any work, education and productivity losses incurred by participants and their carers. The modified version of the TIC-P employed in this study comprise six sections enquiring about health care visits, support received
  - Page 4 of 6 [DRAFT] both at and outside of school, medications and supplements, work, and education and productivity losses incurred by both parents and children.
Treatment Satisfaction Scale | Post-test (week 20)
  The children and parents both will fill this questionnaire. This is a short 6-item parent and adolescents self-report instrument, measuring satisfaction with group attendance. Each item is scored on a 4-point Likert scale with response options ranging from "Yes, very much" to "No" with an open comment section, encouraging participants to freely share their experiences with the intervention.
Change in the Social responsiveness scale - Second Edition (SRS-2) | Baseline (week 0), Post-test (week 20) and follow up (week 36) and long follow up (74 weeks)
  This measure will be used as the parent's primary outcome.The Social Responsiveness Scale - Second Edition (SRS-2) School-Age Form is a 65-item rating scale, designed to measure social deficits in individuals with ASD via parent proxy report has been used as the primary outcome in a previous study evaluating KONTAKT and has been used as the basis for the power calculation for the present RCT. The SRS-2 (2014) enables calculation of a universal score and five treatment subscales: social awareness, social cognition, social communication, social motivation, and restricted interests and repetitive behaviour. These subscales are designed to align closely with the DSM-5 criteria for ASD. The scale takes approximately 15 to 20 minutes to complete with items scored on a 4-point Likert-type scale, ranging from "not true (0)" to "almost always true (3)". The expected value for individuals with a primary diagnosis of ASD is approximately 100.
International classification of functioning (ICF) - Autism coreset | Baseline (week 0), Post-test (week 20) and follow up (week 36) and long follow up (74 weeks)
  evaluates the impact of a disability and its context on an individual's functioning. For the purpose of this study only item related to the KONTAKT© objectives (social communication and interaction) will be selected from the Autism Core set after the manual has been translated to English.
Junior Temperament and characteristic Inventory (JTCI) | Baseline (week 0), Post-test (week 20) and follow up (week 36)
  2.4. This parent-report and child self-report is derived from the International classification of functioning's autism coreset that identifies the personality traits of young children aged 6-16 under 5. Responses are dichotomous (True or False).
Motivation to participate | Weekly through the intervention until post test time from week 1 to 20
  is a weekly measure specifically designed for this study to evaluate the motivation to participate in the groups (both intervention and control) and will be assessed through a 2-item child and parent self-report and a parents proxy-report text, asking "On a scale of 1-5 (as demonstrated by emoji) how much did you like attending this week's group?" and "On a scale of 1-5 (as demonstrated by emoji) how interested are you in attending the next session?" To check for reliability, the results from this measure will be attached to the participants' attendance in the groups.
Change in the LERID friendship questionnaire | Baseline (week 0), Post-test (week 20) and follow up (week 36) and long follow up (74 weeks)
  the LERID friendship questionnaire is a 46-item self-report measure of children's perceptions of the quality of their relationship with their best friend around 11 different aspects of friendship experience: commitment, security, satisfaction, intimacy, protection from victimization, help, affection received from the friend, trust of the friend, trust received from the friend, comfort, Validation and Authenticity of the friendship. The measure is rated on a 5-point Likert scale from "Not true" (1) to "Really true" (5).
Change in the Social Interaction anxiety scale (SIAS) | Weekly through the intervention until post test time from week 1 to 20
  Social Interaction Anxiety Scale (SIAS) is self-report used mainly with adults. The measure has been used with adolescents participating in the KONTAKT program. This study will only use the items which became significant in that study. The measure is scored on a 5-point Likert scale from "Not at all (0)" to "Extremely (4)". The higher scores on the scale indicate higher social interaction anxiety experienced.

CONTACTS AND LOCATIONS:
Locations (1):
- Curtin University, Bentley, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No
Have no ethics to do this

REFERENCES:
- [Derived] Hayden-Evans M, Afsharnejad B, Lee EAL, Milbourn B, Picen T, Johnson M, Bolte S, Girdler S. "I made friends a lot more easily": children and families' experiences of social group programs for children on the autism spectrum. BMC Pediatr. 2025 May 3;25(1):353. doi: 10.1186/s12887-025-05686-6. PMID 40316953
- [Derived] Afsharnejad B, Lee EAL, Hayden-Evans M, Black MH, Alach T, Fridell A, Coco C, Johnson M, Bolte S, Girdler S. Adaptation and Feasibility of KONTAKT Social Skills Toolbox Group Program for Australian Autistic Children. Scand J Child Adolesc Psychiatr Psychol. 2024 Dec 5;12(1):20240011. doi: 10.2478/sjcapp-2024-0011. eCollection 2024 Jan. PMID 39649127